CLINICAL TRIAL: NCT00714831
Title: Referral From Primary Health Care Centers to a Physical Activity Program: Establishing Long-Term Adherence? A Randomized Controlled Trial
Brief Title: Referral From Primary Health Care Centers to a Physical Activity Program. A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Unitat de Suport a la Recerca, Barcelona, Spain (Other); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Maria Giné-Garriga, Primary Health Care of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI081304
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Sedentary General Population
Keywords: Physical activity promotion; Primary health care; Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CG (Active Comparator): Control Group
  Interventions: Behavioral: Health educational program
- IG (Experimental): Intervention Group
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — 3-months physical activity intervention
  Arms: IG
Behavioral: Health educational program — Health education sessions and stretching sessions
  Arms: CG

SUMMARY:
Declining physical activity and the associated rising burden of disease is a major public-health problem and it has long been known that being physically active has positive health effects. The virtual absence of a public health practice infrastructure for the promotion of physical activity at the local level presents a critical challenge to control policy for chronic disease. We aimed to assess the efficacy of a 3-months physical activity program in primary health care to create adherence to physical activity in sedentary individuals.

DETAILED DESCRIPTION:
Physical inactivity has emerged as an important risk factor for many chronic diseases. The decline in physical activity is a key public health concern.

Objective. The objective of the study is to assess the effectiveness of a 3-months physical activity programme in the primary healthcare centres (HC), combined with community resources and interdisciplinary work, to create adherence to physical activity in sedentary individuals.

Methods. The design of the study is a randomized controlled trial with a randomized selection of the sample. A total of 424 subjects of both sexes, older than 18 years old, with a low physical activity level (IPAQ), independent, with no medical contraindication to practice physical activity, and coming from 8 different HC, will participate in the study. Each subject will be offered to participate voluntarily in a physical activity programme (24 sessions, twice a week, 60 minutes/session). There will be two groups of 15-20 subjects in each HC (a total of 8 HC), randomizing the subjects of the intervention (GI) and control groups (GC). The study will be divided in two phases, and in each phase there will be 16 groups (8 GC and 8 GI).

In the first and last session different parameters will be assessed in all the subjects (GC and GI): (1) quality of life related to health with SF-12 questionnaire, (2) the attitude towards practicing physical activity with Prochaska stage changes, (3) the physical activity level with the reduced version of the IPAQ, (4) health perception with COOP/WONCA questionnaire, and (5) the social support for physical activity with SSPAS. The welfare pressure to the HC of each participant is also registered, during the 6 months previous and after the programme. Subjects of GI will go through the 24 sessions while subjects of GC will go through a health educational program and will be asked to continue with their everyday activities. After 3, 6 and 12 months of the end of the programme, a pursuit by means of a call will be done (IPAQ, SF-12 and SSPAS). After 6 and 12 months of the end of the programme the same call will be used to assess the Prochaska stages.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both gender.
* Low physical activity level assessed with International Physical Activity Questionnaire.
* Able to walk and stand up from a chair unaided.

Exclusion Criteria:

* Recommended contradictions to advising physical activity to older adults.
* Presence of unstable angina.
* Uncontrolled congestive heart failure.
* Unstable arrhythmia or heart valvular disease.
* Progressive or debilitating medical conditions.
* Severe hypertension (systolic ≥ 200, or diastolic ≥ 120).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
This randomized controlled trial was designed to assess the effectiveness of a primary care physical activity intervention, in increasing adherence to physical activity in general population, as well as their self-reported physical activity. | baseline-3-6-12-18

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martin, PhD, MD, Study Director — Primary Health Care of Barcelona
Locations (1):
- Primary Health Care, Barcelona, Spain

REFERENCES:
- [Derived] Martin-Borras C, Gine-Garriga M, Puig-Ribera A, Martin C, Sola M, Cuesta-Vargas AI; PPAF Group. A new model of exercise referral scheme in primary care: is the effect on adherence to physical activity sustainable in the long term? A 15-month randomised controlled trial. BMJ Open. 2018 Mar 3;8(3):e017211. doi: 10.1136/bmjopen-2017-017211. PMID 29502081
- [Derived] Gine-Garriga M, Martin-Borras C, Puig-Ribera A, Martin-Cantera C, Sola M, Cuesta-Vargas A; PPAF Group. The Effect of a Physical Activity Program on the Total Number of Primary Care Visits in Inactive Patients: A 15-Month Randomized Controlled Trial. PLoS One. 2013 Jun 21;8(6):e66392. doi: 10.1371/journal.pone.0066392. Print 2013. PMID 23805219
- [Derived] Gine-Garriga M, Martin C, Martin C, Puig-Ribera A, Anton JJ, Guiu A, Cascos A, Ramos R. Referral from primary care to a physical activity programme: establishing long-term adherence? A randomized controlled trial. Rationale and study design. BMC Public Health. 2009 Jan 22;9:31. doi: 10.1186/1471-2458-9-31. PMID 19161605